CLINICAL TRIAL: NCT03465839
Title: The Efficacy of Bedside Nursing Handovers in Improving Information Exchange Quality in Surgical Patients: a Randomised Controlled Trial
Brief Title: Bedside Nursing Handovers in the Surgical Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Piedmont (Other)
Collaborators: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Marco Clari, Adjunct professor, University of Eastern Piedmont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UPO1
Record Dates: First submitted 2018-02-27; First posted 2018-03-14 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: General Surgery
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedside handover (Experimental): Education for improving handovers quality + Education for improving bedside handovers
  Interventions: Behavioral: Education for improving handovers quality; Behavioral: Education for improving bedside handovers
- Control (Active Comparator): Education for improving handovers quality
  Interventions: Behavioral: Education for improving handovers quality

INTERVENTIONS:
Behavioral: Education for improving handovers quality — Specific education on the importance of handovers quality will be provided. The educational session will last 4 hours. The program will be divided into the following sections: 1) a structured survey on the perception of the participants on the handovers importance; 2) Key theoretical concepts on the relevance of handovers with case studies of errors related to this critical moment; 3) showing movie clips of nursing handovers to critically interpret the clips by the participants; 4) presentation of the SBAR method recommended by WHO; 5) general presentation of the nursing delivery assessment project of the Valduce Hospital.
Behavioral: Education for improving bedside handovers — In addition to the education for improving handovers quality, the following intervention will be implemented for nurses assigned to the study department. The course will be supplemented by a section of the duration of an hour, containing 1) information on the principles underlying bedside handovers; 2) how to handle information in front of the patient and on his / her direct involvement; 3) role-playing of the bedside handover will be performed, assigning the roles of nurse and patient among the participants to bring out impressions linked to the functions.
  Arms: Bedside handover

SUMMARY:
Nursing handovers are performed 2-3 times a day for each patient, with an approximate average of 2 million nursing deliveries per year in a hospital of medium size. Nursing handovers are considered essential for the continuity and safety of care. If the relevant clinical information is not shared in a precise and timely manner, it may worsen the patients' outcomes with an increase in adverse events, delays or inappropriate treatment until the omission of procedures.

The modality of nursing delivery presents, therefore, a gap of vulnerability where vital information could not be considered and systematically shared.

Patients should be involved in their care to promote a patient-centred approach. The involvement of patients in handovers is effective compared to other delivery methods.

To date, however, the best mode to deliver handovers was still unclear due to a systematic lack of studies to identify the best practice of nursing handovers. The studies in the literature lack of sound methodologies due to not randomized designs.

Thus an intervention to improve quality of handovers and to implement bedside handovers in surgical wards will be performed.

The following hypotheses were made:

* The introduction of nursing bedside handovers will improve the quality of the information exchanged.
* The educational intervention training intervention will positively modify the nursing handovers.
* There is a relationship between the qualitative level of nursing handovers and working status (expert vs novice) of the nurses.
* There is a relationship between the qualitative level of nursing handovers and the patients' characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients
* All nurses working with surgical patients who attended the educational intervention

Exclusion Criteria:

* Nurses who did not participate in the educational intervention
* Nursed who did not operate stably in the surgical wards included in the study
* New hired nurses

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in handover quality | Baseline, at 1 month after intervention, at 6 months after intervention
  Handoff CEX (Clinical Examination) [3-9 overall on 6 items about setting, organisation, communication, content, judgment, professionalism; 3 worst - 9 best]

SECONDARY OUTCOMES:
Handover length | Baseline, at 1 month after intervention
  Time x handover
Missed care / procedures / diagnostic tests | Baseline, at 1 month after intervention, at 6 months after intervention
  Number of missed care / procedures / diagnostic tests
Patients satisfaction | Baseline, at 1 month after intervention, at 6 months after intervention
  Visual Analogic Scale for satisfaction [0-10; 0 worst - 10 best]

CONTACTS AND LOCATIONS:
Overall Officials: Marco Clari, RN, PhD s, Principal Investigator — University of Eastern Piedmont
Locations (1):
- Valuduce Hospital, Como, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smeulers M, Lucas C, Vermeulen H. Effectiveness of different nursing handover styles for ensuring continuity of information in hospitalised patients. Cochrane Database Syst Rev. 2014 Jun 24;2014(6):CD009979. doi: 10.1002/14651858.CD009979.pub2. PMID 24957503
- [Background] Abraham J, Kannampallil T, Patel VL. A systematic review of the literature on the evaluation of handoff tools: implications for research and practice. J Am Med Inform Assoc. 2014 Jan-Feb;21(1):154-62. doi: 10.1136/amiajnl-2012-001351. Epub 2013 May 23. PMID 23703824
- [Background] Clemow R. Care plans as the main focus of nursing handover: information exchange model. J Clin Nurs. 2006 Nov;15(11):1463-5. doi: 10.1111/j.1365-2702.2006.01524.x. No abstract available. PMID 17038108
- [Background] Chaboyer W, McMurray A, Johnson J, Hardy L, Wallis M, Sylvia Chu FY. Bedside handover: quality improvement strategy to "transform care at the bedside". J Nurs Care Qual. 2009 Apr-Jun;24(2):136-42. doi: 10.1097/01.NCQ.0000347450.90676.d9. PMID 19287252